CLINICAL TRIAL: NCT02269618
Title: Innovative Multidisciplinary Telehealth Program in COPD and CHF Patients: a Randomized Control Trial.
Brief Title: Telehealth Program in Chronic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, Michele Vitacca, Responsible of Respiratory Unit, Fondazione Salvatore Maugeri
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: N.160
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Heart Failure
Keywords: Telehealth, Home-based, rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Group A) (Active Comparator): The patients will be followed in the usual care manner by GPs and by routine specialist visits, if needed
  Interventions: Other: Usual care
- Intervention group (Group B) (Other): Group B (Home-based intervention): the patients will be followed at home for 4 months by nurse and therapist and will perform an individual rehabilitative program. The interventions will be:
  1. Home-based telehealth program
  2. Home-based rehabilitation
  Interventions: Other: Home-based telehealth program; Other: Home-based rehabilitation; Other: Usual care

INTERVENTIONS:
Other: Home-based telehealth program — Home-based telehealth program
  * Scheduled calls initiated by nurse performed weekly; the nurse carried out a standardized interview on general clinical condition of the patients.
  * Unscheduled calls initiated by patients or caregivers through the service centre(24h/24h) to report any clinical problems. in case of signs or symptoms
  * Telemonitoring: during calls, patients can transmit via landline or mobile phone the recordings from the 1-lead ECG to a service centre, and talk to the nurse or doctor
  * Home visit performed by therapist seven days after hospital discharge by setting the daily physical activity and other home visits in case of need
  * Scheduled calls initiated by therapist performed weekly aimed at increasing workload and evaluating the proper execution of exercises.
  Arms: Intervention group (Group B)
Other: Home-based rehabilitation — Home-based rehabilitation Individual rehabilitative program including at least 3 sessions/week of mini-ergometer and exercises and 2 sessions/week of walking with pedometer
  * Mini-ergometer: The personalized protocol will be structured at the beginning on the basis of data obtained from the assessment of the baseline exercise test, trying to get a training activity to the maximum value of around a Borg dyspnoea and motor equal to 6 (according to the protocol of Maltais)
  * Walking: The patient will be encouraged to walk every day. Will be given a pedometer and will be asked to try to increase the amount of steps up to the maximal for the patient.
  Arms: Intervention group (Group B)
Other: Usual care — Usual care All patients will be followed also in usual care manner by their GPs.

SUMMARY:
The aim of this randomized control study is to determine the feasibility and efficacy of an innovative multidisciplinary telehealth program in chronic obstructive pulmonary disease (COPD) and chronic heart failure (CHF) patients. 120 patients (1:1) will be included in the study and followed for 4 months and for additional 2 months of follow-up. The primary outcome is to improve tolerance capacity

DETAILED DESCRIPTION:
COPD and CHF frequently coexist, causing a significant worsening in the quality of life of the patients and increasing morbidity and mortality. The prevalence of COPD in the CHF patients ranges from 20% to 32% of cases, and CHF is prevalent in more than 20% of patients with COPD.

COPD and CHF patients are complicated and frail with a high risk of re-hospitalizations; for this reason an individualized and multidisciplinary program need to be implemented in these patients. The chronic disease trend is fluctuating, burdened by many exacerbations through a vicious circle with dyspnoea, decreased activity, new exacerbations, depression and social isolation, leading to death.

The weight of evidence from a meta-analysis of randomized trials indicates that a multidisciplinary disease-management approach has the best outcomes in terms of prolonged survival and reduced hospital-readmission rates. Home-based management might, arguably, be the preferred approach after hospitalization of chronic diseases patients.

Home-base management might provide an opportunity to prevent clinical deterioration and hospitalizations by a comprehensive, long-term intervention with regular reinforcement of patient adherence, knowledge, and skills. A personalized hospital-discharge programme seems to be the best approach to plan the follow-up care of patients with chronic diseases.

These programmes, particularly important in the care of patients with multiple comorbidities, should include a routine self-management support, consisting in education to recognize symptoms early, to manage medical devices, to identify barriers to adherence to therapy such as adverse effects of drugs, and to check that the intensity of physical therapy is appropriate.

Our study want to investigate feasibility and efficacy of a multidisciplinary telehealth and tele-rehabilitation home based program in patients with COPD and CHF. This is an integrated, multidisciplinary nurse and therapist oriented program; these two figures have a central role during home based intervention and became an essential interface in the dialogue between patient and specialist. The nurse and therapist, each for their competence, collect information, carry out education and training, verify adherence to drug and physical therapy, verify the quality of caregiver assistance. When needed, they require intervention of specialist for consultation or second-opinion.

After drug therapy optimization and physical rehabilitation program definition, the patient will be allocated randomly into 2 groups: 1. Group A (usual care): the patients will be followed in the usual care manner by General Practitioner (GP) and routine specialist visits. 2. Group B (Home-based intervention): the patients will be monitored at home for 4 months by nurse and therapist and they will perform an individual rehabilitative program including at least 3 sessions/week of mini-ergometer and exercises and 2 sessions/week of walking with pedometer.

At baseline, after 4 months and further 2 months of follow-up all patients in both groups will undergo to follows clinical and physical evaluations:

1. ECG (T0; T4 if needed)
2. Echocardiogram (T0, T4 if needed
3. Spirometry (T0 or a spirometry available in the previous year)
4. Arterial blood gases (T0; T4)
5. Walking test (T0; T4; T6)
6. Metabolic Holter monitoring using the Body Monitoring Multi-Sensor Armband (BMSA) (SenseWear) worn at the triceps of the right arm for at least 72 h. (T0; T4; T6)

The questionnaires and scale :

1. Minnesota (T0;T4;T6)
2. COPD Assessment Test (CAT) (T0;T4;T6)
3. Barthel (T0;T4;T6)
4. Dyspnoea and muscle fatigue by Borg scale evaluation, referred by patient during his regular day (T0;T4;T6)
5. Medical Research Council (MRC) scale for dyspnoea during regular day (T0;T4;T6)
6. Physical activity scale for the elderly (PASE) (T0;T4;T6)
7. Customer satisfaction (T4, only group B)

ELIGIBILITY:
Inclusion Criteria:

* COPD new GOLD classification (B, C and D class) and a spirometry in the previous year and
* Systolic and/or diastolic CHF defined at least by an echocardiogram performed in clinical stability; II, III and IV New York Heart Association class and optimized drug therapy.
* Informed consent signed

Exclusion Criteria:

* Physical activity limitations caused by non-cardiac and/or pulmonary problems
* Obstructive Cardiomyopathies and/or myocarditis
* Non cardiac and/or pulmonary pathologies that would cause the death of the patient during the study
* Poor adherence and compliance of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2013-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Improvement tolerance capacity | 4 months and 6 months
  The improvement in tolerance capacity will be measured by walking test performance (meters walked)

SECONDARY OUTCOMES:
Reduction of hospitalisations for cardiovascular disease and /or respiratory disease | 4 months
Reduction of hospitalisations for all-cases | 4 months
energy expenditure and duration and quantification of physical activity Energy expenditure and duration and quantification of physical activity | 4 months and 6 months
  The outcome will be measured in a subgroup of patients using metabolic holter monitoring using the Body Monitoring Multi-Sensor Armband (BMSA) (SenseWear) worn at the triceps of the right arm for at least 72 h.
Improvement of quality of life | 4 months
  The improvement in quality of life, measured by Minnesota Questionnaire and CAT
Reduction of clinical instabilities without hospital admission | 4 months
  The reduction of clinical instabilities will be measured by number of times that patients need to use antibiotics and/or corticosteroids and/or number of times that patients need to increase dosage of diuretic
Reduction of impairment/disability | 4 months
  The reduction of impairment/disability will be measured with Barthel index
Adherence to at least 70% proposal rehabilitative sessions | 4 months and 6 months
  The adherence will be calculated only in the group B

CONTACTS AND LOCATIONS:
Overall Officials: Michele Vitacca, MD, Study Chair — Fondazione Salvatore Maugeri
Locations (3):
- Italy (3):
  - FSM Respiratory Unit, Lumezzane, BS
  - Fondazione Salvatore Maugeri, Cardiology Unit, Lumezzane, BS
  - Fondazione Salvatore Maugeri, Telemedicine Service, Lumezzane, BS

REFERENCES:
- [Background] Hawkins NM, Petrie MC, Jhund PS, Chalmers GW, Dunn FG, McMurray JJ. Heart failure and chronic obstructive pulmonary disease: diagnostic pitfalls and epidemiology. Eur J Heart Fail. 2009 Feb;11(2):130-9. doi: 10.1093/eurjhf/hfn013. PMID 19168510
- [Background] Staszewsky L, Wong M, Masson S, Barlera S, Carretta E, Maggioni AP, Anand IS, Cohn JN, Tognoni G, Latini R; Valsartan Heart Failure Trial Investigators. Clinical, neurohormonal, and inflammatory markers and overall prognostic role of chronic obstructive pulmonary disease in patients with heart failure: data from the Val-HeFT heart failure trial. J Card Fail. 2007 Dec;13(10):797-804. doi: 10.1016/j.cardfail.2007.07.012. PMID 18068611
- [Background] Macchia A, Monte S, Romero M, D'Ettorre A, Tognoni G. The prognostic influence of chronic obstructive pulmonary disease in patients hospitalised for chronic heart failure. Eur J Heart Fail. 2007 Sep;9(9):942-8. doi: 10.1016/j.ejheart.2007.06.004. Epub 2007 Jul 12. PMID 17627878
- [Background] Almagro P, Castro A. Helping COPD patients change health behavior in order to improve their quality of life. Int J Chron Obstruct Pulmon Dis. 2013;8:335-45. doi: 10.2147/COPD.S34211. Epub 2013 Jul 24. PMID 23901267
- [Background] Walters JA, Cameron-Tucker H, Courtney-Pratt H, Nelson M, Robinson A, Scott J, Turner P, Walters EH, Wood-Baker R. Supporting health behaviour change in chronic obstructive pulmonary disease with telephone health-mentoring: insights from a qualitative study. BMC Fam Pract. 2012 Jun 13;13:55. doi: 10.1186/1471-2296-13-55. PMID 22694996
- [Background] Vitacca M, Bianchi L, Guerra A, Fracchia C, Spanevello A, Balbi B, Scalvini S. Tele-assistance in chronic respiratory failure patients: a randomised clinical trial. Eur Respir J. 2009 Feb;33(2):411-8. doi: 10.1183/09031936.00005608. Epub 2008 Sep 17. PMID 18799512
- [Background] Giordano A, Scalvini S, Zanelli E, Corra U, Longobardi GL, Ricci VA, Baiardi P, Glisenti F. Multicenter randomised trial on home-based telemanagement to prevent hospital readmission of patients with chronic heart failure. Int J Cardiol. 2009 Jan 9;131(2):192-9. doi: 10.1016/j.ijcard.2007.10.027. Epub 2008 Jan 28. PMID 18222552
- [Background] Paneroni M, Colombo F, Papalia A, Colitta A, Borghi G, Saleri M, Cabiaglia A, Azzalini E, Vitacca M. Is Telerehabilitation a Safe and Viable Option for Patients with COPD? A Feasibility Study. COPD. 2015 Apr;12(2):217-25. doi: 10.3109/15412555.2014.933794. Epub 2014 Aug 5. PMID 25093419
- [Background] McLean S, Nurmatov U, Liu JL, Pagliari C, Car J, Sheikh A. Telehealthcare for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2011 Jul 6;2011(7):CD007718. doi: 10.1002/14651858.CD007718.pub2. PMID 21735417
- [Background] Shaw RJ, McDuffie JR, Hendrix CC, Edie A, Lindsey-Davis L, Williams JW Jr. Effects of Nurse-Managed Protocols in the Outpatient Management of Adults with Chronic Conditions [Internet]. Washington (DC): Department of Veterans Affairs (US); 2013 Aug. Available from http://www.ncbi.nlm.nih.gov/books/NBK241377/ PMID 25210722
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633
- [Derived] Bernocchi P, Scalvini S, Galli T, Paneroni M, Baratti D, Turla O, La Rovere MT, Volterrani M, Vitacca M. A multidisciplinary telehealth program in patients with combined chronic obstructive pulmonary disease and chronic heart failure: study protocol for a randomized controlled trial. Trials. 2016 Sep 22;17(1):462. doi: 10.1186/s13063-016-1584-x. PMID 27659741